CLINICAL TRIAL: NCT02193997
Title: Double-blind, Placebo-controlled Study to Examine the Effects of Dietary Fiber in Treating Childhood Constipation
Brief Title: Constipation Fiber Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Warren Bishop (Other)
Responsible Party: Sponsor-Investigator, Warren Bishop, MD, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201203734
Record Dates: First submitted 2014-06-24; First posted 2014-07-18 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Functional Constipation in Children
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fiber 1 (Experimental): Fiber bar containing inulin as fiber soucre taken once daily for 4 weeks
  Interventions: Other: Fiber
- Fiber 2 (Experimental): Fiber bar containing soluble corn as fiber soucre taken once daily for 4 weeks
  Interventions: Other: Fiber
- Placebo (Placebo Comparator): Bar with low fiber content (placebo) once daily for 4 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Fiber
  Other Names: Single fiber type
  Arms: Fiber 1
Other: Fiber
  Other Names: Blend of fiber types
  Arms: Fiber 2
Other: Placebo
  Arms: Placebo

SUMMARY:
This study examines the effects of dietary fiber in the treatment of functional childhood constipation.

DETAILED DESCRIPTION:
This is a 4-week double-blind, placebo-controlled study to examine the effects of dietary fiber in treating functional childhood constipation. The addition of fiber is anticipated to allow children to have more normal stool consistency and frequency.

All participants will be asked to take a snack bar twice daily and will be randomized in a 1:1:1 ratio to fiber 1, fiber 2 or placebo snack bar groups. All participants will be asked to take low-dose Miralax to avoid worsening of constipation in all groups.

ELIGIBILITY:
Inclusion Criteria:

* 2-16 years of age with functional constipation as defined based on the Rome III criteria

Exclusion Criteria:

* Constipation attributable to organic and anatomic causes or intake of medication
* Children who had previous surgery of the colon or anus
* History of allergy/intolerance to components of snack bar (e.g. celiac disease)

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in stool frequency | 4 weeks
Change in stool consistency | 4 weeks
  Stool consistency (using the Bristol scale) will be compared between groups, between baseline and study end

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bishop, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States